CLINICAL TRIAL: NCT06298539
Title: The Sensory Attenuation Paradigm in Auditory Modality in Obesity
Brief Title: Auditory Sensory Attenuation in Obesity
Acronym: Ud_SA_OB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 21C308
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: obesity; sensory attenuation; interpersonal difficulties; sense of agency
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: BMI > 30 kg/m2
- Healthy weight: BMI range: 19 - 29 kg/m2

SUMMARY:
The goal of this observational cross-sectional study is to test the sensory attenuation effect with auditory stimuli comparing women with obesity and healthy-weight women. Specifically, the study aims to test whether the sensory attenuation effect (i.e., the perceived loudness of a self-generated sound is weaker than when another person produces the same sound):

i) is observed in obesity ii) it can be modulated in interactive action contexts, as was previously observed in healthy participants.

Participants will compare the loudness of target sound with a comparison tone, which can be prompt by the participant by pressing a button on their own will (i.e., individual context) or upon the experimenter's signal (i.e., interactive context); externally-generated sounds are produced in the opposite way.

DETAILED DESCRIPTION:
The perceived loudness of a self-generated sound is generally weaker than when another person produces the same sound. This effect is known as sensory attenuation, and it is considered a proof of sense of agency (i.e., it relies on the anticipation of the sensory-motor effects of one's intentional action). Recently, it was suggested that this effect is enhanced in interactive action contexts in healthy individuals, meaning that sounds are produced as a consequence of cooperation between individuals.

Participants will compare the loudness of target sound with a comparison tone, which could be generated in 4 different conditions:

i) participants press a button ii) the experimenter press the button iii) participants press the button upon the experimenter's signal (i.e., who touch the participants' arm) iv) the experimenter presses the button upon the participants' signal (i.e., who touch the experimenter's arm).

However, it is not clear whether the same effect of cooperation can be observed also when individuals experience difficulties in social interactions and relationships.

To this purpose, the study compared the sensory attenuation effect for auditory stimuli in a traditional (i.e., individual) and interactive context, comparing women with obesity and healthy-weight women.

Indeed, relational difficulties and social withdrawal characterized this clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2 (controls)
* handedness: right

Exclusion Criteria:

* history of eating disorders (controls)
* major psychiatric conditions (e.g., psychosis, personality disorders)
* developmental disorders (e.g., autism spectrum disorders)
* neurological or brain injuries disorders
* motor impairments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with obesity will be recruited at the IRCCS Istituto Auxologico Italiano, San Giuseppe Hospital, Piancavallo, VB, Italia during their rehabilitative treatment.
  Healthy weight participants will be recruited in the local community and among researchers' contacts.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
point of subjective equality (PSE) | day 1
  individual PSE in each experimental condition is obtained by fitting observed judgements of loudness, relative to seven possible comparison tones. The PSE represents the tone loudness that participants perceive as loud as the target sound (i.e., the sound intensity which records only 50% of correct judgments "which sounds was louder?")

SECONDARY OUTCOMES:
cognitive empathy | day 1
  Interpersonal Reactivity Index - IRI: 28-item self-report questionnaire on a 5-point Likert scale (from 1 -does not describe me well to 5 - describes me very well). Four components of cognitive empathy are measured: i) perspective taking (IRI-PT); ii) fantasy (IRI-F); iii) empathic concern (IRI-EC); iv) personal distress (IRI-PD); each subscale includes 7 items (total scores range from 1 to 35): the higher the score, the higher the expression of cognitive empathy described in each subscale.
interpersonal pleasure | day 1
  Anticipatory and Consummatory Interpersonal Pleasure Scale - ACIPS: 17-item self-reported questionnaire scored on 6-point Likert scale (from 1 - very false for me to 6-very true for me). ACIPS total score ranges from 1 to 102: higher scores indicate higher anticipatory and consummatory interpersonal pleasure.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, San Giuseppe Hospital, Piancavallo, VCO, Italy

IPD SHARING:
Plan to Share IPD: Yes
anonymized experimental raw data
Access Criteria: upon reasonable request to the Authors through the repository platform. Log-in on the platform is required.
URL: https://www.zotero.org/

REFERENCES:
- [Background] Scarpina F, Fossataro C, Sebastiano AR, Bruni F, Scacchi M, Mauro A, Garbarini F. Behavioural evidence of altered sensory attenuation in obesity. Q J Exp Psychol (Hove). 2022 Nov;75(11):2064-2072. doi: 10.1177/17470218211065766. Epub 2021 Dec 29. PMID 34825612
- [Background] Weiss C, Herwig A, Schutz-Bosbach S. The self in social interactions: sensory attenuation of auditory action effects is stronger in interactions with others. PLoS One. 2011;6(7):e22723. doi: 10.1371/journal.pone.0022723. Epub 2011 Jul 27. PMID 21818373